CLINICAL TRIAL: NCT00772733
Title: A Project Ensuring Quality and Cooperation in the Chronic Obstructive Pulmonary Disease (COPD) Treatment
Acronym: KOSMOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn.E.Eriksson, MD, VP Medical, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RDK-DUM-2007/1
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: COPD; Chronic Diseases
Keywords: Quality assurance; rehabilitation; chronic care model; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to ensure the quality of the COPD treatment in primary care by implementing planned follow-up visits, where the disease condition is evaluated and optimised in accordance with the national COPD recommendations. If relevant the general practitioner (GP) will refer patients to COPD rehabilitation conducted by relevant municipality rehabilitation teams. Secondarily the purpose is to improve collaboration and communication between the local hospital pulmonologist, GPs and the municipality rehabilitation team

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnose, verified by spirometry
* Having given informed consent

Exclusion Criteria:

-

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed patients with COPD, verified by spirometry in general practise and/or municipalities.
Sampling Method: Non-Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Control visits at General practitioners | 6-12 months
Lung function measured by spirometry | 6-12 months

SECONDARY OUTCOMES:
Dyspnoea on MRC scale | 6-12 months
Smoking status | 6-12 months
Rehabilitation completed in the municipality rehabilitation team | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Skov Jensen, MD, Study Chair — Region Hospital Viborg, DK; Tina Brandt Sorensen, MD, Study Chair — Region Hospital Horsens, DK; Ove Grann, Principal Investigator — Aalborg
Locations (11):
- Denmark (11):
  - Research Site, Aarhus, Arhus
  - Research Site, Bjerringbro, Viborg
  - Research Site, Møldrup, Viborg
  - Research Site, Skals, Viborg
  - Research Site, Aalborg
  - Research Site, Klarup
  - Research Site, Skive
  - Research Site, Spøttrup
  - Research Site, Stoholm
  - Research Site, Viborg
  - Research Site, Ørum